CLINICAL TRIAL: NCT06458673
Title: Prediction of Growth Trend of Pulmonary Nodules Based on Multi-temporal and Multimodal Medical Data and Its Impact on Pulmonary Nodule Management Strategies
Brief Title: A Prospective, Non-interventional Cohort Study of Subsolid Pulmonary Nodules
Status: Not yet recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Peking University People's Hospital (Other); Guangxi Medical University (Other); Shanghai Zhongshan Hospital (Other); The Third Xiangya Hospital of Central South University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); The Third People's Hospital of Chengdu (Other); Shantou Central Hospital (Other); Hainan Cancer Hospital (Other); Shenzhen People's Hospital (Other); Hunan Cancer Hospital (Other); Shenzhen Third People's Hospital (Other); First Affiliated Hospital of Jinan University (Other); Haikou People's Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Xue-Ning Yang, Vice-Chief of Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital
Other Study IDs: CONAN
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Solitary Lung Nodule; Multiple Pulmonary Nodules
Keywords: Lung Nodule; Prospective; Observational Study
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some studies have shown that the model for judging and predicting the growth of sub-solid pulmonary nodules through big data and deep learning can detect nodule growth earlier. Since most of the training data come from large foreign samples, most of the validated data are CT data from a single center or a few centers, and their generalization ability needs to be further verified. In order to better study subsolid pulmonary nodules in the lungs in China, we plan to conduct a prospective, multicenter, non-interventional observational cohort study.

DETAILED DESCRIPTION:
Through the follow-up of pulmonary nodules, artificial intelligence based on CT was used to study the natural evolution process of subsolid pulmonary nodules, as well as the development law and prognosis of pulmonary subsolid nodules under treatment or no treatment according to clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years old, gender is not limited
* Confirmed subsolid pulmonary nodule by CT, initial pulmonary nodule ≥ 5 mm (including subsolid components) and ≤ 30 mm, do not shrink or disappear after 3 months Follow-up.
* ECOG 0～2
* Able to provide CT in DICOM format
* Informed consent obtained

Exclusion Criteria:

* Long-term use of immunosuppressants and hormone drugs
* History of previous malignancy (if there is no recurrence or carcinoma in situ for more than 5 years after receiving curative therapy, it can be enrolled)
* Inability to cooperate with regular follow-up
* Poor general condition, with the life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subsolid pulmonary nodules of 5 to 30 mm in size found on CT
Sampling Method: Non-Probability Sample
Enrollment: 1184 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
5-year growth rate of subsolid pulmonary nodules | Regular follow-up was carried out according to clinical guidelines and local hospital guidelines, with an interval of 3-6 months and a duration of 5 years
  The 5-year growth rate of the nodules is calculated by comparing the initial and final diameters of the nodules during the follow-up period.Results are expressed as percentages.

SECONDARY OUTCOMES:
Median time from enrollment to invasive diagnosis/intervention in patients with subsolid pulmonary nodules | The time from patient enrollment and initiation of follow-up until invasive diagnosis/intervention
  Median length of time from patient enrollment to invasive diagnosis or therapeutic intervention such as surgical excision, biopsy, or other therapeutic procedures
Lung cancer-specific 5-year survival rate | From the time the patient is enrolled, and follow-up is initiated, up to 5 years of follow-up
  Lung cancer-specific 5-year survival rate is defined as a proportion of patients diagnosed with lung cancer who survive within 5 years of diagnosis
explore the growth rate and pattern of radiographic changes of different types of pulmonary nodules | From the time the patient is enrolled, and follow-up is initiated, up to 5 years of follow-up
  the growth rate is calculated by comparing the initial and final diameters of the nodules during the follow-up period. Results are expressed as 1mm/year
Sensitivity and specificity of radiomics in predicting the growth of subsolid pulmonary nodules | From the time the patient is enrolled, and follow-up is initiated, up to 5 years of follow-up
  the sensitivity and specificity is calculated by comparing the predicted results and the real results

CONTACTS AND LOCATIONS:
Overall Officials: Xuening Yang, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China